CLINICAL TRIAL: NCT02824835
Title: The Effect of the Plant Hormones Strigolactones on Cultures of Dysplastic Colonic Lesions and Cancer
Brief Title: Strigolactones and Dysplastic Colonic Lesions or Cancer
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Meir Medical Center (Other)
Responsible Party: Principal Investigator, ido laish, MD, Meir Medical Center
Other Study IDs: IDO123
Record Dates: First submitted 2016-06-27; First posted 2016-07-07 (Estimated); Last update posted 2016-07-07 (Estimated); Status verified 2016-07

CONDITIONS: Colonic Neoplasms; Colonic Polyps
MeSH Terms: conditions — Colonic Neoplasms; Colonic Polyps

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- adenoma group: Patients with adenoma. Biopsies are taken before endoscopic resection.
  Interventions: Procedure: biopsy during colonoscopy
- cancer group: Patients with colorectal cancer. Biopsies are taken before surgical resection.
  Interventions: Procedure: biopsy during colonoscopy

INTERVENTIONS:
Procedure: biopsy during colonoscopy — sampling the lesion with forcept biopter

SUMMARY:
The purpose of this study is to determine the effects of the plant hormones strigolactones, on cell cultures of colonic polyps and colorectal cancer.

DETAILED DESCRIPTION:
Strigolactones have been shown to anti-proliferative and pro-apoptotic effects in cell cultures of breast and prostate origin, partially by down-regulation of cyclin B1 and induction of cell cycle arrest. In this study the investigators intend to take biopsies from benign colonic polyps and cancer tissue, culture intestinal explants and generate immortalized primary cells as a platform to assess the effect of this plant hormone on cell viability, cell mobility, apoptosis and cytoskeleton modifications.

ELIGIBILITY:
Inclusion Criteria:

* Patients with positive findings during colonoscopy

Exclusion Criteria:

* Patients below 18 years old
* Patients who cannot sign a consent form

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients undergoing colonoscopy who have positive findings (polyps, cancer) during the procedure
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2016-07; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
percentage of cells with reduced viability after dose-dependent exposure | 24 hours of exposure to strigolactone
percentage of cells in G2/M arrest after dose-dependent exposure | 24 hours of exposure to strigolactone
  analysis of cell cycle

CONTACTS AND LOCATIONS:
Overall Officials: Ido Laish, MD, Principal Investigator — Meir Medical Center

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mayzlish-Gati E, Laufer D, Grivas CF, Shaknof J, Sananes A, Bier A, Ben-Harosh S, Belausov E, Johnson MD, Artuso E, Levi O, Genin O, Prandi C, Khalaila I, Pines M, Yarden RI, Kapulnik Y, Koltai H. Strigolactone analogs act as new anti-cancer agents in inhibition of breast cancer in xenograft model. Cancer Biol Ther. 2015;16(11):1682-8. doi: 10.1080/15384047.2015.1070982. Epub 2015 Jul 20. PMID 26192476
- [Background] Pollock CB, Koltai H, Kapulnik Y, Prandi C, Yarden RI. Strigolactones: a novel class of phytohormones that inhibit the growth and survival of breast cancer cells and breast cancer stem-like enriched mammosphere cells. Breast Cancer Res Treat. 2012 Aug;134(3):1041-55. doi: 10.1007/s10549-012-1992-x. Epub 2012 Mar 29. PMID 22476848